CLINICAL TRIAL: NCT04632576
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Sleeping After General Anesthesia in Gynecological Laparoscopic Surgery
Brief Title: Acupoint Stimulation and Postoperative Sleep
Acronym: ASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJH-A-20220325
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia; Sleep
Keywords: anesthetics; sleep; surgery

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- transcutaneous electrical acupoint stimulation (Experimental): transcutaneous electrical acupoint stimulation is one of the many forms of acupuncture, and is a distinctive part of Chinese medicine that has been practiced in China for thousands of years. It is employed by placing electrodes on acupoint and electrical stimulation is given after anesthetic induction to the end of the surgery.
  Interventions: Other: transcutaneous electrical acupoint stimulation
- Control (No Intervention): Electrodes are placed on same acupoints as the experimental group, and will receive the "optimal intensity test" before the anesthesia induction, but no electrical stimulation is given during the operation.

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation — Electrodes will be attached on the surface of acupoints and electrical stimulation will given.
  Other Names: TEAS
  Arms: transcutaneous electrical acupoint stimulation

SUMMARY:
Sleeping model can be affected after surgery. Anesthetics may be involved in the change. The changing of sleeping mode may exert adverse effect on postoperative recovery. Acupuncture and related techniques has been used for treating sleeping disorder. In this study, the effect of transcutaneous electrical acupoint stimulation on sleeping model after general anesthesia will be observed.

DETAILED DESCRIPTION:
Sleep is a necessary, naturally occurring physiologic state that is especially critical to cognition and physical functioning in surgical settings.Poor postoperative sleep is associated with many significant deleterious effects. Therefore, improving overall sleep during postoperative rehabilitation is desirable.

Transcutaneous electrical acupoint stimulation (TEAS) is a non-invasive acupuncture therapy combining the transcutaneous electrical nerve stimulation, and has been utilized in clinical settings for many years. Previous study demonstrated that TEAS combined with anesthesia can upregulate the levels of melatonin and aminobutyric acid to relief central inhibition, thus improve patients'sleep efficiency, prolong total sleep time (TST) and promote sleep quality.

The current study is to examine the effect of perioperative TEAS on subjective and objective sleep quality among patients who have undergone Gynecological laparoscopic surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria

1. Patients scheduled for elective Gynecological laparoscopic surgery under general anesthesia
2. Patients aged 18-65 years
3. Patients with a body mass index (BMI) at 18-30kg/m2
4. Patients with American Society of Anesthesiologists (ASA) grades I-III
5. Patients who provide written informed consent

Exclusion Criteria

1. Participants with sleep apnea or moderate and severe obstructive sleep apnea syndrome (defined by Apnea Hypopnea Index (AHI))
2. Participants with preoperative sleep disturbances (diagnostic criteria of sleep disturbances according to the International Classification of Sleep Disorders, Third Edition (ICSD-3));
3. Participants with central nervous system and mental disease, or difficult to communicate, or unable to cooperate with the investigators.
4. Participants with contraindications to the use of electroacupuncture (including those with infection or injury of the skin to attach electrodes, and those with implanted electronic devices).
5. Participants who had severe diseases of the cardiovascular or hematopoietic systems, or had severe hepatic or renal insufficiency kidney disease
6. Participants with a history of alcohol or drug abuse. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
total sleeping time during the first postoperative night | the first postoperative night
  The primary outcome is the total sleep time on the first postoperative night according to the sleep diary monitored by actigraphy.

SECONDARY OUTCOMES:
Total sleep time during the first 24h after surgery | from discharge from post-anesthesia care unit to 24hours later, totally 24 hours
  total sleep time recorded on the actigraphy on the first perioperative night
the Pittsburgh Sleep Quality Index (PSQI) questionnaire for the last month before surgery | the 1 month before hospitalization
  The PSQI is used to indicate the sleep quality in the last 1 month.
The Athens Insomnia Scale (AIS) score | from discharge from post-anesthesia care unit to 24hours later, totally 24 hours
  The highest score on the Athens Scale is 24, while the lowest score is 0. The higher the score, the more serious the sleep disorder
the Epworth Sleepiness Scale (ESS) score | from discharge from post-anesthesia care unit to 24hours later, totally 24 hours
  ESS scores range from 0 to 24, with higher scores indicating higher levels of sleepiness
the 15-item Quality of Recovery Scale (QoR-15) score | from discharge from post-anesthesia care unit to 24hours later, totally 24 hours
  The QoR-15 score ranges from 0 to 150, and the higher the score, the better the postoperative recovery
Total intraoperative propofol dosage | From the time of anesthetic induction to the end of the surgery
  the total dosage used for the anesthetic induction and maintenance
Times for the needs of rescue analgesics | from discharge from operation room to 24 hours later, totally 24 hours
  Times for the needs of rescue analgesics in the first 24h.
Number of episodes of postoperative adverse events | from discharge from the operation room to 48 hours later, totally 48 hours
  Number of episodes of postoperative adverse events such as nausea and vomiting, delirium, pulmonary edema, septic shock, arrhythmia, etc after surgery.
time of intestinal recovery after surgery | from discharge from the operation room to 48 hours later, totally 48 hours
  time to first flatus, time to food intake, catheter remove and ambulation
length of postoperative hospital stay | from date of randamization until the time of discharge from the hospital from any cause,assessed up to 5 days
  length of postoperative hospital stay
total wake time during the first 24h after surgery | from discharge from post-anesthesia care unit to 24hours later, totally 24 hours]
  recorded on the actigraphy on the first perioperative night

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Northwest Women's and Children's Hospital, Xi'an, Shaanxi
  - the First Affiliated Hospital of the Air Force Military Medical University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Xi 'an Hospital of Traditional Chinese Medicine, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Individual data including protocol and statistical analysis plan will be shared during 3 months and 5 years following article publication after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: during 3 months and 5 years following article publication after deidentification

REFERENCES:
- [Background] Song B, Chang Y, Li Y, Zhu J. Effects of Transcutaneous Electrical Acupoint Stimulation on the Postoperative Sleep Quality and Pain of Patients After Video-Assisted Thoracoscopic Surgery: A Prospective, Randomized Controlled Trial. Nat Sci Sleep. 2020 Oct 27;12:809-819. doi: 10.2147/NSS.S270739. eCollection 2020. PMID 33154688